CLINICAL TRIAL: NCT07394257
Title: Intrastromal Moxifloxacin as an Adjunctive Therapy in Recalcitrant Bacterial Keratitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan, lecturer of ophthalmology, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1827
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bacterial Keratitis; Recalcitrant Infectious Keratitis; Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed using a computer-generated random sequence. Allocation will be concealed using sealed opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrastromal moxifloxacin injection plus standard topical moxifloxacin therapy (Experimental): Intrastromal injection of preservative-free moxifloxacin 0.5% using a 30-gauge needle under aseptic conditions.
  Interventions: Drug: Intrastromal moxifloxacin injection plus standard topical moxifloxacin therapy
- Standard topical moxifloxacin therapy alone (Experimental): • Intensive topical moxifloxacin eye drops every 1-2 hours initially, tapered according to standard clinical protocol and response
  Interventions: Drug: Standard topical moxifloxacin therapy alone

INTERVENTIONS:
Drug: Intrastromal moxifloxacin injection plus standard topical moxifloxacin therapy — Intrastromal injection of preservative-free moxifloxacin 0.5% using a 30-gauge needle under aseptic conditions.
  Arms: Intrastromal moxifloxacin injection plus standard topical moxifloxacin therapy
Drug: Standard topical moxifloxacin therapy alone — Intensive topical moxifloxacin eye drops every 1-2 hours initially, tapered according to standard clinical protocol and response.
  Arms: Standard topical moxifloxacin therapy alone

SUMMARY:
Bacterial keratitis is a potentially sight-threatening corneal infection that is commonly treated with intensive topical antibiotics. Despite appropriate therapy, some cases show inadequate clinical response, particularly when the infection involves the deep corneal stroma. Limited penetration of topical antibiotics into deeper corneal layers may contribute to treatment failure in these recalcitrant cases.

Intrastromal antibiotic injection is a targeted drug-delivery approach that allows high local antimicrobial concentrations directly at the site of infection. Moxifloxacin is a broad-spectrum fluoroquinolone with proven efficacy in bacterial keratitis and favorable corneal tissue penetration. However, evidence regarding the clinical benefit and safety of intrastromal moxifloxacin as an adjunctive treatment remains limited.

This randomized controlled trial aims to evaluate the efficacy and safety of intrastromal moxifloxacin injection as an adjunct to standard topical moxifloxacin therapy compared with topical therapy alone in patients with recalcitrant bacterial keratitis. The primary outcome is time to complete clinical resolution of infection. Secondary outcomes include visual acuity improvement, ulcer healing rate, need for additional interventions, and treatment-related complications.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * Clinical diagnosis of bacterial keratitis confirmed by corneal scraping and microbiology
  * Recalcitrant keratitis defined as no significant clinical improvement after 48-72 hours of intensive topical antibiotic therapy
  * Ability to provide written informed consent

Exclusion Criteria

* Fungal, viral, or acanthamoeba keratitis
* Corneal perforation or impending perforation
* Known hypersensitivity to fluoroquinolones
* Pregnancy or lactation
* Immunocompromised state or current systemic immunosuppressive therapy
* Previous intrastromal or intracameral antibiotic injection for the same episode

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete clinical resolution(days) | weekly till complete healing
  Time to complete clinical resolution, defined as corneal re-epithelialization with disappearance of stromal infiltrate and anterior chamber reaction.

SECONDARY OUTCOMES:
• Epithelial defect size(mm) | weekly for one month
  epithelial defect is measured by surgical caliper
Hypopyon height(mm). | weekly for one month
Pain score on visual Analog scale (VAS, 1 - 10). | weekly for one month
Best-corrected visual acuity (BCVA) (LogMAR or Snellen) | weekly for one month
Complications (perforation, thinning, endophthalmitis). | after 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Ramadan Amer, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
(IPD) will not be shared because the study was not designed with a data-sharing framework, and participants did not provide explicit consent for secondary use or external sharing of their individual-level data. In addition, sharing IPD may pose potential risks to participant privacy, even after de-identification, particularly in single-center studies with limited sample sizes. Current clinical trial registration requirements mandate transparency regarding data-sharing intentions but do not obligate investigators to share IPD. Therefore, the decision not to share IPD is made in accordance with ethical standards, privacy regulations, and applicable registry policies.

REFERENCES:
- [Background] Zemba M, et al. Intrastromal injections in infectious keratitis. Pharmaceutics. 2023
- See also: Related Info — https://doi.org/10.1016/j.ophtha.2006.12.011